CLINICAL TRIAL: NCT00537329
Title: A Phase IIIB Pilot Study Of Efficacy And Safety Of Anidulafungin In The Treatment Of Candidemia In Asian Patients
Brief Title: Anidulafungin In Treatment Of Candidemia In Asian Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A8851016; PF-03910960
Record Dates: First submitted 2007-09-25; First posted 2007-10-01 (Estimated); Results first posted 2010-02-17 (Estimated); Last update posted 2010-03-09 (Estimated); Status verified 2010-03

CONDITIONS: Candidemia
MeSH Terms: conditions — Candidemia | interventions — Anidulafungin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Open (Other): This is an open-label, multi-center, non-comparative 12 week study evaluating the efficacy and safety of anidulafungin in subjects with candidemia.
  Interventions: Drug: Anidulafungin

INTERVENTIONS:
Drug: Anidulafungin — Eligible subjects will be initiated on a single loading dose of 200 mg IV anidulafungin, followed by 100 mg IV anidulafungin once daily for a minimum of 5 days but not more than 42 days.

SUMMARY:
The purpose of this study is to determine whether or not the Investigational Study Drug anidulafungin is safe and effective in the treatment of a fungal infection, candidemia, in Asian subjects.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with at least one positive blood test for Candida pathogen from a blood sample taken within 96 hours prior to start of study treatment.
* Subjects with clinical evidence of candida infection within 48 hours prior to enrollment.
* Acute Physiology and Chronic Health Enquiry (APACHE) score less than or equal to 20.

Exclusion Criteria:

* Prior exposure to systemic antifungals for more than 48 hours.
* Subjects who had, at any time, previously received anidulafungin.
* Subjects with poor venous (vein) access that would inhibit the administration of the intravenous study drug or withdrawing of multiple blood samples.
* Life expectancy < 72 hours.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2008-01; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (13):
- India (5):
  - Pfizer Investigational Site, Ahmedabad, Gujarat
  - Pfizer Investigational Site, Bangalore, Karnataka
  - Pfizer Investigational Site, Mumbai, Maharashtra
  - Pfizer Investigational Site, Ludhiana, Punjab
  - Pfizer Investigational Site, Noida, Uttar Pradesh
- Pfizer Investigational Site, Legaspi Village, Makati City, Philippines
- Taiwan (4):
  - Pfizer Investigational Site, Banqiao District, Taipei
  - Pfizer Investigational Site, Taichung
  - Pfizer Investigational Site, Tainan
  - Pfizer Investigational Site, Taipei
- Thailand (3):
  - Pfizer Investigational Site, Pathumwan, Bangkok
  - Pfizer Investigational Site, Amphoe Mueang, Changwat Khon Kaen
  - Pfizer Investigational Site, Amphoe Mueang, Chiang Mai

REFERENCES:
- [Derived] De Rosa FG, Busca A, Capparella MR, Yan JL, Aram JA. Invasive Candidiasis in Patients with Solid Tumors Treated with Anidulafungin: A Post Hoc Analysis of Efficacy and Safety of Six Pooled Studies. Clin Drug Investig. 2021 Jun;41(6):539-548. doi: 10.1007/s40261-021-01024-7. Epub 2021 Apr 23. PMID 33891293
- [Derived] Sganga G, Wang M, Capparella MR, Tawadrous M, Yan JL, Aram JA, Montravers P. Evaluation of anidulafungin in the treatment of intra-abdominal candidiasis: a pooled analysis of patient-level data from 5 prospective studies. Eur J Clin Microbiol Infect Dis. 2019 Oct;38(10):1849-1856. doi: 10.1007/s10096-019-03617-9. Epub 2019 Jul 6. PMID 31280481
- [Derived] Kontoyiannis DP, Bassetti M, Nucci M, Capparella MR, Yan JL, Aram J, Hogan PA. Anidulafungin for the treatment of candidaemia caused by Candida parapsilosis: Analysis of pooled data from six prospective clinical studies. Mycoses. 2017 Oct;60(10):663-667. doi: 10.1111/myc.12641. Epub 2017 Jun 9. PMID 28597967
- [Derived] Kullberg BJ, Vasquez J, Mootsikapun P, Nucci M, Paiva JA, Garbino J, Yan JL, Aram J, Capparella MR, Conte U, Schlamm H, Swanson R, Herbrecht R. Efficacy of anidulafungin in 539 patients with invasive candidiasis: a patient-level pooled analysis of six clinical trials. J Antimicrob Chemother. 2017 Aug 1;72(8):2368-2377. doi: 10.1093/jac/dkx116. PMID 28459966
- [Derived] Mootsikapun P, Hsueh PR, Talwar D, Co VM, Rajadhyaksha V, Ong ML. Intravenous anidulafungin followed optionally by oral voriconazole for the treatment of candidemia in Asian patients: results from an open-label Phase III trial. BMC Infect Dis. 2013 May 15;13:219. doi: 10.1186/1471-2334-13-219. PMID 23676114
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A8851016&StudyName=Anidulafungin%20In%20Treatment%20Of%20%20Candidemia%20In%20Asian%20Subjects

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Approximately 100 eligible subjects from 22 centers were planned to be enrolled. However, due to slow enrollment, 46 subjects were screened and 43 subjects were assigned to treatment.
Groups:
- Anidulafungin: Single 200 milligram (mg) intravenous (IV) dose of anidulafungin, followed by anidulafungin 100 mg IV once daily (QD) for a minimum of 5 days but not more than 42 days.
Period: Overall Study
Arm/Group | Anidulafungin
Started | 43
Completed | 17
Not Completed | 26
Not completed — Death | 10
Not completed — Adverse Event | 3
Not completed — Lack of Efficacy | 2
Not completed — Lost to Follow-up | 6
Not completed — Withdrawal by Subject | 4
Not completed — Other | 1

BASELINE CHARACTERISTICS:
Arm/Group | Anidulafungin
Number analyzed (Participants) | 43
Age, Customized [Number; unit: participants]
  Between 18 and 44 years | 10
  Between 45 and 64 years | 15
  ≥ 65 years | 18
Age Continuous [Mean (Standard Deviation); unit: years] | 56.5 (18.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 23

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Global Response of Success at End of Treatment
Description: Number of subjects with clinician assessed global response of success; defined as cure (resolution of signs and symptoms of Candida infection) or improvement (significant but incomplete resolution of signs and symptoms of Candida infection) on the clinical response in conjunction with eradication (follow up negative culture result for Candida species [spp]) or presumed eradication (follow up culture was not available and clinical outcome defined as success) on the microbiological response.
Time Frame: End of treatment (EOT) = Day 5 up to Day 42
Population: Modified Intent to Treat (MITT): includes all Full Analysis Set (FAS) subjects (received at least 1 dose of study treatment) with confirmed, documented diagnosis of candidemia and had received the initial loading dose of study treatment.
Measure: Number; unit: participants
Arm/Group | Anidulafungin
Number analyzed (Participants) | 42
participants | 31
Statistical Analysis 1: Comparison: Anidulafungin; Sample size enrollment of 100 subjects was planned. Assuming an overall response rate of 75 percent (%), a 95% confidence interval (CI) for the percentage of subjects responding to treatment would have ranged from 66.3% to 83.7% allowing for 5% nonevaluability. This would have provided a level of precision considered acceptable for this Asian regional study; Test type: Superiority or Other; 2-sided exact Clopper-Pearson (percent) = 86.1, 95% CI [70.5 to 95.3]

2. Secondary Outcome: Number of Subjects With Global Response of Success at Endpoints
Description: Number of subjects with clinician assessed global response of success. Defined as cure or improvement (cure/improvement): cure=resolution of signs and symptoms of Candida infection; improvement=significant but incomplete resolution of signs and symptoms of Candida infection on the clinical response in conjunction with eradication or presumed eradication (erad/presumed erad): erad=follow up negative culture result for Candida spp; presumed erad=follow up culture was not available and clinical outcome defined as success on the microbiological response.
Time Frame: End of intravenous treatment (EOIT), end of Week 2 after EOT (2 Wks post EOT), end of Week 6 after EOT (6 Wks post EOT), at end of 12 weeks after baseline (12 Wks post baseline)
Population: MITT; EOT visit could occur anytime from Day 5 through Day 42; if a subject terminated early, the timeframe "at end of 12 weeks after baseline" could occur in the follow-up period (6 Wks post EOT or Week 12 post EOT).
Measure: Number; unit: participants
Arm/Group | Anidulafungin
Number analyzed (Participants) | 42
participants
  EOIT | 33
  2 Wks post EOT | 24
  6 Wks post EOT | 17
  12 Wks post baseline | 16
Statistical Analysis 1: Comparison: Anidulafungin; EOIT; Test type: Superiority or Other; 2-sided exact Clopper-Pearson (percent) = 89.2, 95% CI [74.6 to 97.0]
Statistical Analysis 2: Comparison: Anidulafungin; 2 Wks post EOT; Test type: Superiority or Other; 2-sided exact Clopper-Pearson (percent) = 82.8, 95% CI [64.2 to 94.2]
Statistical Analysis 3: Comparison: Anidulafungin; 6 Wks post EOT; Test type: Superiority or Other; 2-sided exact Clopper-Pearson (percent) = 89.5, 95% CI [66.9 to 98.7]
Statistical Analysis 4: Comparison: Anidulafungin; 12 Wks post baseline; Test type: Superiority or Other; 2-sided exact Clopper-Pearson (percent) = 72.7, 95% CI [49.8 to 89.3]

3. Secondary Outcome: Number of Subjects With Clinical Response of Success at Endpoints
Description: Number of subjects with clinician assessed clinical response (CR) of success. Defined as cure or improvement (cure/improvement): cure=resolution of signs and symptoms of Candida infection; improvement=significant but incomplete resolution of signs and symptoms of Candida infection on the clinical response.
Time Frame: EOIT, EOT (Day 5 up to Day 42), 2 Wks post EOT, 6 Wks post EOT, 12 Wks post baseline
Population: MITT. EOT visit could occur anytime from Day 5 through Day 42; if a subject terminated early, the timeframe "at end of 12 weeks after baseline" could occur in the follow-up period (6 Wks post EOT or Week 12 post EOT).
Measure: Number; unit: participants
Arm/Group | Anidulafungin
Number analyzed (Participants) | 42
participants
  EOIT: success (cure/improvement) | 34
  EOIT: cure | 27
  EOIT: improvement | 7
  EOT: success (cure/improvement) | 32
  EOT: cure | 27
  EOT: improvement | 5
  2 Wks post EOT: success (cure/improvement) | 26
  2 Wks post EOT: cure | 25
  2 Wks post EOT: improvement | 1
  6 Wks post EOT: success (cure/improvement) | 17
  6 Wks post EOT: cure | 16
  6 Wks post EOT: improvement | 1
  12 Wks post baseline: success (cure/improvement) | 17
  12 Wks post baseline: cure | 17
  12 Wks post baseline: improvement | 0
Statistical Analysis 1: Comparison: Anidulafungin; EOIT: success (cure/improvement); Test type: Superiority or Other; 2-sided exact Clopper-Pearson (percent) = 97.1, 95% CI [85.1 to 99.9]
Statistical Analysis 2: Comparison: Anidulafungin; EOT: success (cure/improvement); Test type: Superiority or Other; 2-sided exact Clopper-Pearson (percent) = 94.1, 95% CI [80.3 to 99.3]
Statistical Analysis 3: Comparison: Anidulafungin; 2 Wks post EOT: success (cure/improvement); Test type: Superiority or Other; 2-sided exact Clopper-Pearson (percent) = 92.9, 95% CI [76.5 to 99.1]
Statistical Analysis 4: Comparison: Anidulafungin; 6 Wks post EOT: success (cure/improvement); Test type: Superiority or Other; 2-sided exact Clopper-Pearson (percent) = 94.4, 95% CI [72.7 to 99.9]
Statistical Analysis 5: Comparison: Anidulafungin; 12 Wks post baseline: success (cure/improvement); Test type: Superiority or Other; 2-sided exact Clopper-Pearson (percent) = 85.0, 95% CI [62.1 to 96.8]

4. Secondary Outcome: Number of Subjects With Microbiological Response of Success at Endpoints
Description: Number of subjects with clinician assessed microbiological response (MR) of success. Defined as eradication or presumed eradication (erad/presumed erad): erad=follow up negative culture result for Candida spp; presumed eradication=follow up culture was not available and clinical outcome defined as success on the microbiological response.
Time Frame: EOIT, EOT (Day 5 up to Day 42), 2 Wks post EOT, 6 Wks post EOT, 12 Wks post baseline
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Anidulafungin
Number analyzed (Participants) | 42
participants
  EOIT: success (erad/presumed erad) | 36
  EOIT: erad | 31
  EOIT: presumed erad | 5
  EOT: success (erad/presumed erad) | 34
  EOT: erad | 31
  EOT: presumed erad | 3
  2 Wks post EOT: success (erad/presumed erad) | 25
  2 Wks post EOT: erad | 22
  2 Wks post EOT: presumed erad | 3
  6 Wks post EOT: success (erad/presumed erad) | 17
  6 Wks post EOT: erad | 14
  6 Wks post EOT: presumed erad | 3
  12 Wks post baseline: success (erad/presumed erad) | 16
  12 Wks post baseline: erad | 14
  12 Wks post baseline: presumed erad | 2
Statistical Analysis 1: Comparison: Anidulafungin; EOIT: success (erad/presumed erad); Test type: Superiority or Other; 2-sided exact Clopper-Pearson (percent) = 97.3, 95% CI [85.8 to 99.9]
Statistical Analysis 2: Comparison: Anidulafungin; EOT: success (erad/presumed erad); Test type: Superiority or Other; 2-sided exact Clopper-Pearson (percent) = 97.1, 95% CI [85.1 to 99.9]
Statistical Analysis 3: Comparison: Anidulafungin; 2 Wks post EOT: success (erad/presumed erad); Test type: Superiority or Other; 2-sided exact Clopper-Pearson (percent) = 86.2, 95% CI [68.3 to 96.1]
Statistical Analysis 4: Comparison: Anidulafungin; 6 Wks post EOT: success (erad/presumed erad); Test type: Superiority or Other; 2-sided exact Clopper-Pearson (percent) = 94.4, 95% CI [72.7 to 99.9]
Statistical Analysis 5: Comparison: Anidulafungin; 12 Wks post baseline: success (erad/presumed erad); Test type: Superiority or Other; 2-sided exact Clopper-Pearson (percent) = 84.2, 95% CI [60.4 to 96.6]

5. Secondary Outcome: Time to Death From Any Cause
Description: Time to death (median survival time in days) from any cause; time to death includes the first day (Day 1) of study drug (baseline and Day 1 allowed to occur on same day). EOT visit could occur anytime from Day 5 through Day 42; if a subject terminated early, the timeframe "at end of 12 weeks after baseline" could occur in the follow-up period (6 Wks post EOT or Week 12 post EOT).
Time Frame: Baseline through end of 12 weeks after baseline
Population: MITT; time to death (median survival time in days) based on Kaplan-Meier method if estimable. Data not summarized by median survival time as planned as median time is not estimable; < 50% of subjects died out of the analyzable population.
Measure: Median (Full Range); unit: days
Arm/Group | Anidulafungin
Number analyzed (Participants) | 0

6. Secondary Outcome: Time to Death Due to Candidemia
Description: Time to death (median survival time in days) due to candidemia; time to death includes the first day (Day 1) of study drug (baseline and Day 1 allowed to occur on same day). EOT visit could occur anytime from Day 5 through Day 42; if a subject terminated early, the timeframe "at end of 12 weeks after baseline" could occur in the follow-up period (6 Wks post EOT or Week 12 post EOT).
Time Frame: Baseline through end of 12 weeks after baseline
Population: MITT; time to death (median survival time in days) based on Kaplan-Meier method if estimable. Data not summarized by median survival time as planned as median time is not estimable; no subjects died due to candidemia out of the analyzable population.
Measure: Median (Full Range); unit: days
Arm/Group | Anidulafungin
Number analyzed (Participants) | 0

7. Secondary Outcome: Absolute Values for β-D-glucan Assay Results at Endpoints in Relation to Clinical Response Status of Success or Status of Failure at End of All Treatment
Description: Absolute values for β-D-glucan (range 0 to 6000 picograms per milliliter [pg/mL]) summarized at all timeframe endpoints by subject's at end of all treatment clinical response status of success (Success at EOT) or failure (Failure at EOT) and as combined status of all subjects (All at EOT). Success: cure (resolution of signs and symptoms of Candida infection) or improvement (significant but incomplete resolution of signs and symptoms); failure: no significant improvement in signs and symptoms or death due to Candida infection; subjects must have received at least 3 doses of anidulafungin.
Time Frame: Baseline, Day 3, Day 5, Day 7, EOT (Day 5 up to Day 42)
Population: MITT; (n)=number of subjects with analyzable data at observation; summary includes only subjects who completed visit; missing or indeterminate CR treated as failures. Failures were carried forward for subjects who withdrew prematurely from study with a documented failure. "All" category includes all subjects with success or failure at EOT.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Anidulafungin
Number analyzed (Participants) | 42
pg/mL
  Success at EOT: baseline β-D-glucan (n=30) | 1095.8 (968.52)
  Failure at EOT: baseline β-D-glucan (n=10) | 1447.9 (2178.27)
  All at EOT: baseline β-D-glucan (n=40) | 1183.9 (1347.71)
  Success at EOT: Day 3 β-D-glucan (n=32) | 1132.0 (1249.22)
  Failure at EOT: Day 3 β-D-glucan (n=4) | 2753.3 (3991.50)
  All at EOT: Day 3 β-D-glucan (n=36) | 1312.1 (1736.33)
  Success at EOT: Day 5 β-D-glucan (n=29) | 1140.5 (1149.22)
  Failure at EOT: Day 5 β-D-glucan (n=6) | 2443.8 (3987.38)
  All at EOT: Day 5 β-D-glucan (n=35) | 1363.9 (1916.80)
  Success at EOT: Day 7 β-D-glucan (n=24) | 1190.8 (1011.93)
  Failure at EOT: Day 7 β-D-glucan (n=4) | 3140.8 (4436.99)
  All at EOT: Day 7 β-D-glucan (n=28) | 1469.4 (1882.17)
  Success at EOT: EOT β-D-glucan (n=28) | 1018.9 (783.76)
  Failure at EOT: EOT β-D-glucan (n=3) | 2917.7 (4737.50)
  All at EOT: EOT β-D-glucan (n=31) | 1202.7 (1541.02)

8. Secondary Outcome: Change From Baseline for β-D-glucan Assay Results at Endpoints in Relation to Clinical Response Status of Success or Status of Failure at End of All Treatment
Description: Change from baseline for β-D-glucan (range 0 to 6000 pg/mL) summarized at endpoints by subject's at end of all treatment clinical response status of Success at EOT or Failure at EOT and as combined status of All at EOT. Success=cure (resolution of signs, symptoms of Candida infection) or improvement (significant but incomplete resolution of signs, symptoms); failure=no significant improvement or death due to Candida infection; subject must have received at least 3 doses of anidulafungin. Percent change calculated as ([mean value of β-D-glucan at observation-baseline value]/baseline value*100).
Time Frame: Baseline, Day 3, Day 5, Day 7, EOT (Day 5 up to Day 42)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Anidulafungin
Number analyzed (Participants) | 42
percent change
  Success at EOT: Day 3 β-D-glucan (n=30) | -0.4 (50.56)
  Failure at EOT: Day 3 β-D-glucan (n=4) | -11.0 (51.50)
  All at EOT: Day 3 β-D-glucan (n=34) | -1.7 (49.99)
  Success at EOT: Day 5 β-D-glucan (n=27) | -1.0 (52.14)
  Failure at EOT: Day 5 β-D-glucan (n=6) | 1.3 (54.36)
  All at EOT: Day 5 β-D-glucan (n=33) | -0.6 (51.68)
  Success at EOT: Day 7 β-D-glucan (n=23) | 4.3 (55.37)
  Failure at EOT: Day 7 β-D-glucan (n=4) | 4.5 (24.14)
  All at EOT: Day 7 β-D-glucan (n=27) | 4.3 (51.59)
  Success at EOT: EOT β-D-glucan (n=27) | 7.0 (69.64)
  Failure at EOT: EOT β-D-glucan (n=3) | 14.0 (18.41)
  All at EOT: EOT β-D-glucan (n=30) | 7.7 (66.15)

9. Secondary Outcome: Absolute Values for β-D-glucan Assay Results at Endpoints in Relation to Microbiological Response Status of Success or Status of Failure at End of All Treatment
Description: Absolute values for β-D-glucan (range 0 to 6000 pg/mL) summarized at timeframe endpoints by subject's at end of all treatment microbiological response status of Success at EOT or Failure at EOT and as combined status of All at EOT. Success: eradication (follow up negative culture for Candida spp) or presumed eradication (follow up culture was not available and clinical outcome defined as success); failure: persistence (follow up culture was positive for at least 1 baseline Candida spp) or presumed persistence (follow up culture was not available and clinical outcome was defined as failure).
Time Frame: Baseline, Day 3, Day 5, Day 7, EOT (Day 5 up to Day 42)
Population: MITT; (n)=number of subjects with analyzable data at observation; summary includes only subjects who completed visit; missing microbiological responses treated as failures. Failures carried forward for subjects who withdrew prematurely from study with documented failure. "All" category includes all subjects with success or failure at EOT.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Anidulafungin
Number analyzed (Participants) | 42
pg/mL
  Success at EOT: baseline β-D-glucan (n=32) | 1219.7 (1491.27)
  Failure at EOT: baseline β-D-glucan (n=8) | 1040.4 (491.35)
  All at EOT: baseline β-D-glucan (n=40) | 1183.9 (1347.71)
  Success at EOT: Day 3 β-D-glucan (n=32) | 1349.0 (1826.61)
  Failure at EOT: Day 3 β-D-glucan (n=4) | 1017.4 (752.22)
  All at EOT: Day 3 β-D-glucan (n=36) | 1312.1 (1736.33)
  Success at EOT: Day 5 β-D-glucan (n=29) | 1444.3 (2087.84)
  Failure at EOT: Day 5 β-D-glucan (n=6) | 975.3 (595.29)
  All at EOT: Day 5 β-D-glucan (n=35) | 1363.9 (1916.80)
  Success at EOT: Day 7 β-D-glucan (n=24) | 1527.2 (2023.77)
  Failure at EOT: Day 7 β-D-glucan (n=4) | 1122.3 (544.01)
  All at EOT: Day 7 β-D-glucan (n=28) | 1469.4 (1882.17)
  Success at EOT: EOT β-D-glucan (n=31) | 1202.7 (1541.02)
  All at EOT: EOT β-D-glucan (n=31) | 1202.7 (1541.02)

10. Secondary Outcome: Change From Baseline for β-D-glucan Assay Results at Endpoints in Relation to Microbiological Response of Status of Success or Status of Failure at EOT
Description: Change from baseline in β-D-glucan (range 0 to 6000 pg/mL) summarized at endpoints and by subject's EOT microbiological response status of Success at EOT or Failure at EOT and as combined status of All at EOT. Success=eradication (negative culture Candida spp or presumed eradication (culture not available, clinical outcome defined as success); failure=persistence (culture positive for at least 1 baseline Candida spp) or presumed persistence (culture not available, clinical outcome defined as failure). Percent change=([mean value of β-D-glucan at observation-baseline value]/baseline value*100).
Time Frame: Baseline, Day 3, Day 5, Day 7, EOT (Day 5 up to Day 42)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Anidulafungin
Number analyzed (Participants) | 42
percent change
  Success at EOT: Day 3 β-D-glucan (n=30) | 0.0 (50.64)
  Failure at EOT: Day 3 β-D-glucan (n=4) | -14.3 (49.60)
  All at EOT: Day 3 β-D-glucan (n=34) | -1.7 (49.99)
  Success at EOT: Day 5 β-D-glucan (n=27) | 0.4 (52.75)
  Failure at EOT: Day 5 β-D-glucan (n=6) | -5.2 (50.95)
  All at EOT: Day 5 β-D-glucan (n=33) | -0.6 (51.68)
  Success at EOT: Day 7 β-D-glucan (n=23) | 5.6 (55.63)
  Failure at EOT: Day 7 β-D-glucan (n=4) | -3.0 (16.97)
  All at EOT: Day 7 β-D-glucan (n=27) | 4.3 (51.59)
  Success at EOT: EOT β-D-glucan (n=30) | 7.7 (66.15)
  All at EOT: Day 7 β-D-glucan (n=30) | 7.7 (66.15)

11. Secondary Outcome: Number of Subjects With Global Response of Success at EOT in Relation to Subject Subgroups
Description: Number of subjects with clinician assessed global response of success at EOT (clinical=cure, improvement, microbiological=eradication, presumed eradication) in relation to subject subgroups (subject may be represented in >1 subgroup). Subgroups: Neutropenic status (absolute neutrophil count [ANC in cubic millimeters [cmm]); baseline pathogen; previous surgery (any surgery, abdominal surgery); organ transplantation (kidney, liver, heart); elderly; renal insufficiency (calculated creatinine clearance [CCC] in milliliters per minute [mL/min]); central venous catheter; receiving chemotherapy.
Time Frame: EOT (Day 5 up to Day 42)
Population: MITT. May have >1 baseline pathogen; previous surgery=any surgery (includes abdominal surgery) within 1 month prior to baseline (PTB); chemotherapy for solid cell tumors or hematological malignancies at baseline or within 3 months PTB; central venous catheter (CVC) up to 1 month PTB; (n)=subjects per subgroup with analyzable data at observation.
Measure: Number; unit: participants
Arm/Group | Anidulafungin
Number analyzed (Participants) | 42
participants
  Neutropenic status: ANC ≤ 500/cmm (n=2) | 1
  Neutropenic status: ANC >500/cmm (n=37) | 28
  Baseline pathogen: Candida albicans (n=14) | 10
  Baseline pathogen: Candida glabrata (n=6) | 4
  Baseline pathogen: Candida parapsilosis (n=4) | 4
  Baseline pathogen: Candida rugosa (n=1) | 1
  Baseline pathogen: Candida tropicalis (n=18) | 13
  Previous surgery: Any surgery (n=13) | 11
  Previous surgery: Abdominal surgery (n=8) | 7
  Elderly: Age ≥ 65 years (n=17) | 10
  Renal insufficiency (CCC < 30 mL/min) (n=11) | 6
  Use of Central venous catheter = Yes (n=21) | 17
  Receiving chemotherapy = Yes (n=7) | 5
Statistical Analysis 1: Comparison: Anidulafungin; Neutropenic status: ANC ≤ 500/cmm; Test type: Superiority or Other; 2-sided exact Clopper-Pearson (percent) = 50.0, 95% CI [1.3 to 98.7]
Statistical Analysis 2: Comparison: Anidulafungin; Neutropenic status: ANC > 500/cmm; Test type: Superiority or Other; 2-sided exact Clopper-Pearson (percent) = 75.7, 95% CI [58.8 to 88.2]
Statistical Analysis 3: Comparison: Anidulafungin; Baseline pathogen: Candida albicans; Test type: Superiority or Other; 2-sided exact Clopper-Pearson (percent) = 71.4, 95% CI [41.9 to 91.6]
Statistical Analysis 4: Comparison: Anidulafungin; Baseline pathogen: Candida glabrata; Test type: Superiority or Other; 2-sided exact Clopper-Pearson (percent) = 66.7, 95% CI [22.3 to 95.7]
Statistical Analysis 5: Comparison: Anidulafungin; Baseline pathogen: Candida parapsilosis; Test type: Superiority or Other; 2-sided exact Clopper-Pearson (percent) = 100.0, 95% CI [39.8 to 100.0]
Statistical Analysis 6: Comparison: Anidulafungin; Baseline pathogen: Candida rugosa; Test type: Superiority or Other; 2-sided exact Clopper-Pearson (percent) = 100.0, 95% CI [2.5 to 100.0]
Statistical Analysis 7: Comparison: Anidulafungin; Baseline pathogen: Candida tropicalis; Test type: Superiority or Other; 2-sided exact Clopper-Pearson (percent) = 72.2, 95% CI [46.5 to 90.3]
Statistical Analysis 8: Comparison: Anidulafungin; Previous surgery: Any surgery; Test type: Superiority or Other; 2-sided exact Clopper-Pearson (percent) = 84.6, 95% CI [54.6 to 98.1]
Statistical Analysis 9: Comparison: Anidulafungin; Previous surgery: Abdominal surgery; Test type: Superiority or Other; 2-sided exact Clopper-Pearson (percent) = 87.5, 95% CI [47.3 to 99.7]
Statistical Analysis 10: Comparison: Anidulafungin; Elderly: Age ≥ 65 years; Test type: Superiority or Other; 2-sided exact Clopper-Pearson (percent) = 58.8, 95% CI [32.9 to 81.6]
Statistical Analysis 11: Comparison: Anidulafungin; Renal insufficiency (CCC < 30 mL/min); Test type: Superiority or Other; 2-sided exact Clopper-Pearson (percent) = 54.5, 95% CI [23.4 to 83.3]
Statistical Analysis 12: Comparison: Anidulafungin; Use of Central venous catheter = Yes; Test type: Superiority or Other; 2-sided exact Clopper-Pearson (percent) = 81.0, 95% CI [58.1 to 94.6]
Statistical Analysis 13: Comparison: Anidulafungin; Receiving chemotherapy = Yes; Test type: Superiority or Other; 2-sided exact Clopper-Pearson (percent) = 71.4, 95% CI [29.0 to 96.3]

ADVERSE EVENTS:
Arm/Group | Anidulafungin
Serious Adverse Events (participants affected / at risk) | 16/43
Other Adverse Events (participants affected / at risk) | 30/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Anidulafungin (N=43)
Cardiac failure congestive (Cardiac disorders) | 1
Cardio-respiratory arrest (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Chills (General disorders) | 1
Pyrexia (General disorders) | 1
Bacteraemia (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Septic shock (Infections and infestations) | 2
Systemic candida (Infections and infestations) | 1
Hypernatraemia (Metabolism and nutrition disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Hypotension (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Anidulafungin (N=43)
Leukopenia (Blood and lymphatic system disorders) | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Acute coronary syndrome (Cardiac disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 2
Asthenopia (Eye disorders) | 1
Conjunctivitis (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Ascites (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 3
Diarrhoea (Gastrointestinal disorders) | 8
Flatulence (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Peritonitis (Gastrointestinal disorders) | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 3
Chest discomfort (General disorders) | 1
Chest pain (General disorders) | 1
Oedema peripheral (General disorders) | 2
Pain (General disorders) | 2
Pitting oedema (General disorders) | 2
Pyrexia (General disorders) | 1
Thirst (General disorders) | 1
Jaundice (Hepatobiliary disorders) | 1
Drug hypersensitivity (Immune system disorders) | 1
Abscess limb (Infections and infestations) | 1
Acarodermatitis (Infections and infestations) | 1
Bacteraemia (Infections and infestations) | 2
Bacterial sepsis (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 1
Nosocomial infection (Infections and infestations) | 1
Oral candidiasis (Infections and infestations) | 3
Pneumonia (Infections and infestations) | 1
Sepsis (Infections and infestations) | 2
Systemic candida (Infections and infestations) | 1
Urosepsis (Infections and infestations) | 1
ECG signs of myocardial ischaemia (Investigations) | 1
Transaminases increased (Investigations) | 1
Cachexia (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Fluid overload (Metabolism and nutrition disorders) | 2
Hyperammonaemia (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 2
Hypernatraemia (Metabolism and nutrition disorders) | 3
Hypocalcaemia (Metabolism and nutrition disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 5
Hypophosphataemia (Metabolism and nutrition disorders) | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Convulsion (Nervous system disorders) | 1
Depressed level of consciousness (Nervous system disorders) | 1
Hepatic encephalopathy (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 2
Confusional state (Psychiatric disorders) | 1
Delirium (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 4
Azotaemia (Renal and urinary disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Hydronephrosis (Renal and urinary disorders) | 1
Renal failure acute (Renal and urinary disorders) | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 2
Choking (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory tract haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 3
Rash pruritic (Skin and subcutaneous tissue disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
Hypertension (Vascular disorders) | 1
Hypotension (Vascular disorders) | 3
Thrombophlebitis (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of < 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), < 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.